CLINICAL TRIAL: NCT02586545
Title: Shared Care for Patients With Type 2 Diabetes Across the Primary and Secondary Health Care Sector
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: Metropolitan University College (Other)
Responsible Party: Principal Investigator, Lene Munch, MHS, Ph.D.-student, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DIA-1234
Record Dates: First submitted 2015-10-21; First posted 2015-10-26 (Estimated); Last update posted 2019-01-03 (Actual); Status verified 2019-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Shared care model (Experimental): Four visits a year: one annual comprehensive check-up at the outpatient diabetes clinic and three quarterly visits at the general practitioner.
  Interventions: Other: Shared care
- Mono sectorial care (No Intervention): Treament as usual including four visits a year with the diabetes team at the outpatient clinic: an annual comprehensive check-up, identical to the one received by the intervention group, and three quarterly visits.

INTERVENTIONS:
Other: Shared care
  Arms: Shared care model

SUMMARY:
The aim of the study is to test the effect of a new shared care model for type 2 diabetes care and compare it with a standardized care management program in a specialized hospital-based out-patient clinic.

The hypothesis is that participants with type 2 diabetes followed in a shared care program will have a comparable outcome in HbA1c to participants receiving standard care.

DETAILED DESCRIPTION:
The prevalence of patients with type 2 diabetes is in growth globally. In order to secure high quality in diabetes care it is necessary to rethink the way in which the care is organized. The investigators want to test a new model of shared care across the interface of primary and secondary care sector for patients with type 2 diabetes who are at risk stratification level 2. Based on a national and regional risk stratification model patients can be stratified to three levels according to risk and complexity of treatment: level 1 (uncomplicated), level 2 (intermediate risk) and level 3 (high risk).

The objective of the study is to show equal outcomes among the participants being treated in either a shared care program or an established program in a specialized outpatient clinic.

The study is a non-inferiority randomized controlled trial. The shared care model will be tested during a period of three years. All participants are offered four medical visits a year. The shared care intervention consists of one annual comprehensive check-up at the outpatient clinic and three quarterly visits at a general practice. The control group is followed with four quarterly visits at the outpatient clinic including an annual comprehensive check-up. The recruitment period spans over approximately 12 months, and participants are randomized to intervention or control group in a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* Must be over the age of 18 years
* The diagnosis of type 2 diabetes
* Risk stratification level 2
* Capable of speaking and writing in Danish
* Give oral and written consent before entering the study

Exclusion Criteria:

* Diagnosed with other types of diabetes than type 2 diabetes
* Risk stratification level 1 or 3
* Being pregnant or breastfeeding
* Having severe co-morbidity with life expectancy less than five years
* Being under such conditions, that the patient will not be able to show up or go through with the appointments (e.g. moderate to severe dementia and severe psychiatric conditions)
* Participating in long-lasting interventions (>2 weeks) that potentially affects the primary outcome in our study or patients participating in studies which include blood sampling amounting to >5 % of the blood volume two months prior to the randomisation and/or the follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline Hemoglobin A, Glycosylated (HbA1c) at 12, 24 and 36 months | Baseline and follow-up at 12, 24 and 36 months

SECONDARY OUTCOMES:
The proportion of patients who meet national standard indicators reflecting quality of care | Follow-up at 12, 24 and 36 months after baseline
  These indicators cover seven areas: HbA1c, blood pressure, low density lipoprotein, albuminuria, fundoscopy, foot examination and smoking status.

OTHER OUTCOMES:
Change from baseline Quality of life at 12, 24 and 36 months | Baseline and follow-up at 12, 24 and 36 months
  Measured by the Short Form 36 (SF-36)
Change from baseline blood pressure at 12, 24 and 36 months | Baseline and follow-up at 12, 24 and 36 months
Change from baseline diabetes symptoms at 12, 24 and 36 months | Baseline and follow-up at 12, 24 and 36 months
  Meassured by the Diabetes Symptom Checklist-revised (DSC-r).

CONTACTS AND LOCATIONS:
Overall Officials: Lene Munch, MHS, Ph.D.-student, Principal Investigator — Center for Diabetes Research, Gentofte Hospital, University of Copenhagen, Denmark. Institute of Nursing, University College Metropol, Denmark.
Locations (1):
- Center for Diabetes Research, Gentofte Hospital, University of Copenhagen, Hellerup, Denmark

REFERENCES:
- [Derived] Munch L, Bennich B, Arreskov AB, Overgaard D, Konradsen H, Knop FK, Vilsboll T, Roder ME. Shared care management of patients with type 2 diabetes across the primary and secondary healthcare sectors: study protocol for a randomised controlled trial. Trials. 2016 Jun 4;17(1):277. doi: 10.1186/s13063-016-1409-y. PMID 27259669